CLINICAL TRIAL: NCT01668589
Title: Prospective Observational Study to Evaluate Medication-taking Behavior With Denosumab (Prolia) and Patient Characteristics in Postmenopausal Women With Osteoporosis in Routine Clinical Practice in Germany, Austria, Greece and Belgium
Brief Title: Observational Study of Denosumab (Prolia®) in Postmenopausal Women With Osteoporosis
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20110126
Record Dates: First submitted 2012-08-16; First posted 2012-08-20 (Estimated); Results first posted 2016-09-20 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Postmenopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The main objective of this observational study was to describe medication-taking behavior of patients treated with denosumab for postmenopausal osteoporosis (PMO) at 12 and 24 months.

DETAILED DESCRIPTION:
The decision to treat patients with denosumab was made independent of and before their enrolment in the study. No study drug was administered as part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Indicated for treatment of osteoporosis in postmenopausal women at increased risk of fractures according to the approved Regional Prescribing Information (eg, EU SmPC in Germany, Austria, Greece and Belgium).
* Enrolled into the study within 4 weeks of receiving their first injection of Prolia® according to the approved Regional Prescribing Information (eg, EU SmPC in Germany, Austria, Greece and Belgium).
* Appropriate written informed consent has been obtained (as required per local country regulations).

Exclusion Criteria:

* Patient is currently enrolled in or has been enrolled within the prior 6 months in a study involving any investigational procedure, device or drug.
* Contraindicated for treatment with Prolia® according to the approved Regional Prescribing Information (eg, EU SmPC in Germany, Austria, Greece and Belgium).
* Participation in ongoing or previous denosumab clinical trials.
* Patient has any kind of disorder that, in the opinion of the investigator, may compromise the ability of the patient to give written informed consent.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Postmenopausal women indicated for treatment of osteoporosis at increased risk of fractures according to the approval regional prescribing information, e.g. EU SmPC
Sampling Method: Non-Probability Sample
Enrollment: 1501 (Actual)
Dates: Start 2011-11-28 (Actual); Primary Completion 2015-08-31 (Actual); Study Completion 2015-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (111):
- Austria (10):
  - Research Site, Graz
  - Research Site, Klagenfurt
  - Research Site, Landeck
  - Research Site, Leibnitz, Styria
  - Research Site, Lieboch
  - Research Site, Salzburg
  - Research Site, Sankt Stefan
  - Research Site, Vienna
  - Research Site, Voitsberg
  - Research Site, Vöcklabruck
- Belgium (47):
  - Research Site, Aalst
  - Research Site, Aarschot
  - Research Site, Alsemberg
  - Research Site, Baisy-Thy
  - Research Site, Blankenberge
  - Research Site, Bornem
  - Research Site, Brain-Le-Comte
  - Research Site, Bruges
  - Research Site, Brussels
  - Research Site, ChÃªnÃ©e
  - Research Site, Dour
  - Research Site, Eisden Maasmechelen
  - Research Site, Genk
  - Research Site, Ghent
  - Research Site, Gribomont
  - Research Site, Grimbergen
  - Research Site, Haine-Saint-Paul
  - Research Site, Halen
  - Research Site, Ham
  - Research Site, Ham-sur-Heure
  - Research Site, Harelbeke
  - Research Site, Hasselt
  - Research Site, Heusden
  - Research Site, Heusy
  - Research Site, Hoeilaart
  - Research Site, Knokke-Heist
  - Research Site, Kortrijk
  - Research Site, Kraainem
  - Research Site, Landen
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Lummen
  - Research Site, Marchovelette
  - Research Site, Mont-Godinne
  - Research Site, Mont-sur-Marchienne
  - Research Site, Mouscron
  - Research Site, Natoye
  - Research Site, Paal-Beringen
  - Research Site, Retie
  - Research Site, Seraing
  - Research Site, Steenokkerzeel
  - Research Site, Stoumont
  - Research Site, Thuilles
  - Research Site, Tongeren
  - Research Site, Vilvoorde
  - Research Site, Vlijtingen-Riemst
  - Research Site, Wetteren
- Germany (45):
  - Research Site, Aachen
  - Research Site, Augsburg
  - Research Site, Bad Kreuznach
  - Research Site, Bad Reichenhall
  - Research Site, Bammental
  - Research Site, Bautzen
  - Research Site, Berlin
  - Research Site, Cottbus
  - Research Site, DÃ¼sseldorf
  - Research Site, Dresden
  - Research Site, Erfurt
  - Research Site, Erlangen
  - Research Site, Freiburg im Breisgau
  - Research Site, Freudenstadt
  - Research Site, Friedrichroda
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Hattingen
  - Research Site, Heidelberg
  - Research Site, Heinsberg
  - Research Site, Herne
  - Research Site, Hettstedt
  - Research Site, Hildesheim
  - Research Site, Immenstadt im Allgäu
  - Research Site, Lahnstein
  - Research Site, Leipzig
  - Research Site, Leverkusen
  - Research Site, Marburg
  - Research Site, MÃ¼llheim
  - Research Site, MÃ¼nchen
  - Research Site, MÃ¼nster
  - Research Site, MÃ¶nchengladbach-Rheydt
  - Research Site, NÃ¼rnbrecht
  - Research Site, Neustadt
  - Research Site, Nienburg
  - Research Site, OsnabrÃ¼ck
  - Research Site, Potsdam
  - Research Site, SaarbrÃ¼cken
  - Research Site, Stockach
  - Research Site, Ulm
  - Research Site, VÃ¶lklingen
  - Research Site, Wadgassen
  - Research Site, WÃ¼rzburg
  - Research Site, Wittstock
  - Research Site, Zerbst
- Greece (9):
  - Research Site, Athens
  - Research Site, Chaidari, Athens
  - Research Site, Chania, Crete
  - Research Site, Heraklion
  - Research Site, Heraklion, Crete
  - Research Site, Livadeia
  - Research Site, Maroussi, Athens
  - Research Site, Pátrai
  - Research Site, Thessaloniki

REFERENCES:
- [Background] Fahrleitner-Pammer A, Papaioannou N, Gielen E, Feudjo Tepie M, Toffis C, Frieling I, Geusens P, Makras P, Boschitsch E, Callens J, Anastasilakis AD, Niedhart C, Resch H, Kalouche-Khalil L, Hadji P. Factors associated with high 24-month persistence with denosumab: results of a real-world, non-interventional study of women with postmenopausal osteoporosis in Germany, Austria, Greece, and Belgium. Arch Osteoporos. 2017 Dec;12(1):58. doi: 10.1007/s11657-017-0351-2. Epub 2017 Jun 22. PMID 28643265
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at various study centers in Germany, Austria, Greece, and Belgium. The recruitment period was from 28 November 2012 to 31 August 2013.
Groups:
- Germany: Participants in Germany who received denosumab 60 mg once every 6 months subcutaneously according to the approved prescribing information for the treatment of postmenopausal osteoporosis (PMO) in routine clinical practice.
- Austria: Participants in Austria who received denosumab 60 mg once every 6 months subcutaneously according to the approved prescribing information for the treatment of postmenopausal osteoporosis (PMO) in routine clinical practice.
- Greece: Participants in Greece who received denosumab 60 mg once every 6 months subcutaneously according to the approved prescribing information for the treatment of postmenopausal osteoporosis (PMO) in routine clinical practice.
- Belgium: Participants in Belgium who received denosumab 60 mg once every 6 months subcutaneously according to the approved prescribing information for the treatment of postmenopausal osteoporosis (PMO) in routine clinical practice.
Period: Overall Study
Arm/Group | Germany | Austria | Greece | Belgium
Started | 600 | 300 | 300 | 301
Received Denosumab | 599 | 300 | 300 | 301
Completed | 461 | 242 | 265 | 266
Not Completed | 139 | 58 | 35 | 35
Not completed — Lost to Follow-up | 29 | 37 | 15 | 5
Not completed — Full Consent/Agreement Withdrawn | 54 | 8 | 11 | 4
Not completed — Death | 12 | 3 | 2 | 11
Not completed — Other | 44 | 10 | 7 | 15

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS), defined as all enrolled patients with enrollment date into the electronic trial operations system, provided informed consent, and received 1 pre-enrollment denosumab injection.
Groups:
- Total: Total of all reporting groups
Arm/Group | Germany | Austria | Greece | Belgium | Total
Number analyzed (Participants) | 579 | 300 | 299 | 301 | 1479
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.5 (8.7) | 71.0 (9.5) | 66.3 (9.2) | 71.2 (10.4) | 70.7 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 579 | 300 | 299 | 301 | 1479
  Male | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Persistent With Denosumab Injections at 12 Months and 24 Months
Description: A participant was considered persistent with denosumab at 12 months if they received at least 1 denosumab injection following the pre-enrolment denosumab injection no later than 6 months + 8 weeks (ie, no greater than 239 days apart).
  A participant was considered persistent with denosumab at 24 months if they received at least 3 denosumab injections following the pre-enrolment denosumab injection, and the length of time between any 2 consecutive denosumab injections did not exceed 6 months + 8 weeks (ie, no greater than 239 days apart).
Time Frame: 12 months and 24 months
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Germany | Austria | Greece | Belgium
Number analyzed (Participants) | 579 | 300 | 299 | 301
percentage of participants
  12 Months | 92.2 [89.7 to 94.3] | 89.3 [85.3 to 92.6] | 94.3 [91.1 to 96.7] | 95.7 [92.7 to 97.7]
  24 Months | 75.1 [71.4 to 78.6] | 79.7 [74.7 to 84.1] | 82.6 [77.8 to 86.7] | 86.0 [81.6 to 89.8]

2. Primary Outcome: Percentage of Participants Adherent to Denosumab Injection at 12 Months and 24 Months
Description: A participant was considered adherent to denosumab at 12 months if they received at least 1 denosumab injection over the 12-month period following the pre-enrolment denosumab injection, with the time between any 2 consecutive injections being at most 6 months ± 4 weeks (between 155 and 211 days apart).
  A participant was considered adherent to denosumab at 24 months if they received at least 3 denosumab injections over the 24-month period following the pre-enrolment denosumab injection, with the time between any 2 consecutive injections being at most 6 months ± 4 weeks (between 155 and 211 days apart).
Time Frame: 12 months and 24 months
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Germany | Austria | Greece | Belgium
Number analyzed (Participants) | 579 | 300 | 299 | 301
percentage of participants
  12 Months | 87.6 [84.6 to 90.1] | 85.0 [80.4 to 88.8] | 89.6 [85.6 to 92.8] | 89.0 [84.9 to 92.3]
  24 Months | 62.9 [58.8 to 66.8] | 66.0 [60.3 to 71.3] | 69.6 [64.0 to 74.7] | 70.1 [64.6 to 75.2]

3. Primary Outcome: Medication Coverage Ratio (MCR) for Denosumab Injection at 12 Months and 24 Months
Description: MCR at 12 months was defined as the accumulative number of days covered with denosumab treatment during the first 12 months divided by 366 days, expressed as a percentage.
  MCR at 24 months was defined as the accumulative number of days covered with denosumab treatment during the first 24 months divided by 732 days, expressed as a percentage.
  It was assumed that each injection of denosumab treatment provided 6 months of coverage (or 183 days) from the date of injection or until the date of the next injection, whichever comes first. So, a participant who received only 1 injection in the first year would have MCR at 12 months equal to 50%.
Time Frame: From baseline to 12 months and 24 months
Population: Full analysis set
Measure: Mean (95% Confidence Interval); unit: percentage of days of coverage
Arm/Group | Germany | Austria | Greece | Belgium
Number analyzed (Participants) | 579 | 300 | 299 | 301
percentage of days of coverage
  12 Months | 94.5 [93.5 to 95.5] | 93.2 [91.6 to 94.9] | 95.8 [94.6 to 96.9] | 96.2 [95.1 to 97.3]
  24 Months | 87.4 [85.8 to 89.1] | 87.9 [85.3 to 90.4] | 91.2 [89.3 to 93.1] | 92.4 [90.5 to 94.2]

4. Secondary Outcome: Time to Non-persistence With Denosumab Injection
Description: Time to non-persistence for non-persistent patients was calculated as the time between the date of the first denosumab injection and the date of last denosumab injection received during the period where the patient was still classified as persistent, plus 6 months (183 days). Participants were considered persistent at 24 months if they received at least 4 injections, including the baseline injection, with no more than 6 months + 8 weeks apart between any 2 consecutive injections.
Time Frame: 24 months
Population: Full analysis set who were non-persistent at 24 months
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Germany | Austria | Greece | Belgium
Number analyzed (Participants) | 144 | 61 | 52 | 42
months | 12.23 [6.03 to 17.89] | 6.03 [6.03 to 13.05] | 12.00 [6.03 to 13.38] | 12.20 [6.03 to 17.51]

5. Secondary Outcome: Percentage of Participants Who Received Denosumab Injections Within the Specified Window
Description: The percentage of participants who received 0, 1, 2, or 3 denosumab injections within the specified window (defined by the persistence definition as 6 months + 8 weeks). The number of injections that a participant took during the 2-year period after the first pre-enrolment injection, and that were given within the appropriate window from the previous injection, irrespective of when the previous injection was given. Only the first 3 post-baseline injections are considered.
Time Frame: 24 months
Population: Full analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Germany | Austria | Greece | Belgium
Number analyzed (Participants) | 579 | 300 | 299 | 301
percentage of participants
  No post-baseline injections | 5.9 (0.9) [6.03 to 17.89] | 9.7 (0.9) [6.03 to 13.05] | 2.7 (0.7) [6.03 to 13.38] | 3.7 (0.7) [6.03 to 17.51]
  1 post-baseline injection | 7.8 | 3.7 | 7.0 | 3.0
  2 post-baseline injections | 11.2 | 7.0 | 7.7 | 7.3
  3 post-baseline injections | 75.1 | 79.7 | 82.6 | 86.0

6. Secondary Outcome: Percent Change From Baseline in Total Hip Bone Mineral Density (BMD) at 24 Months
Description: Bone mineral density was measured using dual energy X-ray absorptiometry (DXA).
Time Frame: Baseline and Month 24
Population: Full analysis set with a baseline value and a month 24 value measured with the same machine type.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Germany | Austria | Greece | Belgium
Number analyzed (Participants) | 100 | 28 | 10 | 31
percent change | 4.4 (6.2) | 4.1 (3.2) | 6.6 (6.6) | 4.1 (6.3)

7. Secondary Outcome: Percent Change From Baseline in Femoral Neck Bone Mineral Density (BMD) at 24 Months
Description: Bone mineral density was measured using dual energy X-ray absorptiometry (DXA).
Time Frame: Baseline and Month 24
Population: Full analysis set with a baseline value and a month 24 value measured with the same body side and machine type.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Germany | Austria | Greece | Belgium
Number analyzed (Participants) | 116 | 28 | 29 | 31
percent change | 3.4 (5.4) | 3.7 (5.7) | 6.0 (9.5) | 3.1 (9.3)

8. Secondary Outcome: Percent Change From Baseline in Lumbar Spine Bone Mineral Density (BMD) at 24 Months
Description: Bone mineral density was measured using dual energy X-ray absorptiometry (DXA).
Time Frame: Baseline and Month 24
Population: Full analysis set with a baseline value and a month 24 value measured with the same machine type.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Germany | Austria | Greece | Belgium
Number analyzed (Participants) | 131 | 24 | 57 | 34
percent change | 6.5 (6.2) | 8.2 (4.6) | 8.4 (8.3) | 7.8 (5.9)

ADVERSE EVENTS:
Time Frame: 24 months
Description: Only adverse drug reactions were collected in this observational study. Serious Adverse Events summarizes serious adverse drug reactions, defined as serious adverse events that are considered related to denosumab.
  Other Adverse Events summarizes the non-serious occurrences of adverse drug reactions that exceeded a 1% frequency threshold.
Groups:
- Germany; Austria; Greece; Belgium: Prolia 60 mg SC Q6M
Arm/Group | Germany | Austria | Greece | Belgium
Serious Adverse Events (participants affected / at risk) | 2/579 | 0/300 | 0/300 | 1/301
Other Adverse Events (participants affected / at risk) | 0/579 | 0/300 | 0/300 | 0/301
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Germany (N=579) | Austria (N=300) | Greece (N=300) | Belgium (N=301)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.